CLINICAL TRIAL: NCT04730388
Title: Evaluation of the Efficacy and Tolerance of the Association ATEZOLIZUMAB - BEVACIZUMAB in the Treatment of a Locally Advanced Hepatocellular Carcinoma Inoperable or Metastatic in Finistère
Brief Title: ATEZOLIZUMAB - BEVACIZUMAB in the Treatment Hepatocellular Carcinoma Inoperable or
Acronym: HEPATOFIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0325
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: ATEZOLIZUMAB, BEVACIZUMAB , Advanced hepatocellular carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the efficacy and safety of the combination ATEZOLIZUMAB - BEVACIZUMAB in the treatment of locally advanced inoperable or metastatic hepatocellular carcinoma in Finistère

DETAILED DESCRIPTION:
Patients treated by ATEZOLIZUMAB and BEVACIZUMAB for an Advanced hepatocellular carcinoma will be followed to observed their safety and the efficacy of this treatment, and to identify prongnosis factors

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma locally advanced or metastatic, non able to be resectable, with no prior systemic treatment
* Child Pugh A and ECOG 0 or 1
* upper digestiuve endoscopy less than 6 months, if esophageal varcices : must be treated
* non eligible to receive a locoregional therpay or progressive after this kinf of treatment
* with informed consent

Exclusion Criteria:

* refuse to participate
* under legal protection
* exclusion criteria from the tempory utilisation authorization

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma locally advanced or metastatic in first line of systemic treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-18 (Estimated); Primary Completion 2022-01-18 (Estimated); Study Completion 2022-01-18 (Estimated)

PRIMARY OUTCOMES:
predictive factor for progression-free survival | 12 months
  progression-free survival = time between treatment initiation and rediologic or clinical progression